CLINICAL TRIAL: NCT04775160
Title: Smartphone-based Ecological Momentary Intervention for Secondary Prevention of Suicidal Thoughts and Behavior: a Randomised Clinical Trial
Brief Title: Smartphone-based Ecological Momentary Intervention for Suicide Prevention: a Randomised Clinical Trial
Acronym: SmartCrisis2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Centre Hospitalier Régional Universitaire Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC005-21_FJD
Record Dates: First submitted 2021-02-21; First posted 2021-03-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will be monitored using smartphone-based active and passive Ecological Momentary Assessment through the MEmind and eB2 mobile applications, and will receive treatment as usual, which will consist of psychiatric follow-up (scheduled appointments with their psychiatrist) in an outpatient Secondary Suicide Prevention Programme, with predetermined clinical reviews according to the Brief Intervention Contact recommendations (1, 2, 4, 7 and 11 weeks, and 4, 6, 9 and 12 months)
- Intervention group (Experimental): The intervention group will receive an Ecological Momentary Intervention called SmartSafe, will be monitored using smartphone-based active and passive Ecological Momentary Assessment through the MEmind and eB2 mobile applications, and their treatment as usual, which will consist of psychiatric follow-up (scheduled appointments with their psychiatrist) in an outpatient Secondary Suicide Prevention Programme, with predetermined clinical reviews according to the Brief Intervention Contact recommendations (1, 2, 4, 7 and 11 weeks, and 4, 6, 9 and 12 months)
  Interventions: Device: SmartSafe

INTERVENTIONS:
Device: SmartSafe — The SmartSafe Ecological Momentary Intervention is contained in the MEmind smartphone application and consists of a Safety plan, an Enhanced contact via app (app-EC) intervention, and a "mental toolbox". The Safety plan is a set of personalized coping strategies that the patient can use in a suicidal crisis. Our safety plan was adapted to a digital environment, including the possibility to activate pre-recorded messages, lead to websites with health resources, or put the patient in contact with the emergency services. The Enhanced contact via app (app-EC) intervention is inspired by the SIAM project and consists in messages that will be sent via the MEmind app inquiring patients about their mental well-being and informing them of the means to request preferential or urgent care. The mental toolbox contains videos relaxation techniques videos and behavioral activation and mentalization exercises.
  Other Names: The SmartSafe Ecological Momentary Intervention
  Arms: Intervention group

SUMMARY:
Introduction: Suicide is one of the leading public health issues worldwide. Mobile health can help us to combat suicide through monitoring and treatment. The SmartCrisis 2.0 randomized clinical trial aims to evaluate the effectiveness of a smartphone-based Ecological Momentary Intervention to prevent suicidal thoughts and behaviour.

Methods and analysis: The SmartCrisis 2.0 study is a randomized clinical trial with two parallel groups, conducted among patients with a history of suicidal behaviour treated at the University Hospital Fundación Jiménez Díaz. The intervention group will be monitored using Ecological Momentary Assessment and will receive an Ecological Momentary Intervention called 'SmartSafe' in addition to their treatment as usual (TAU). TAU will consist of psychiatric follow-up of the patient (scheduled appointments with a psychiatrist) in our outpatient Suicide Prevention clinic, with predetermined clinical appointments according to the Brief Intervention Contact recommendations (1, 2, 4, 7 and 11 weeks, and 4, 6, 9 and 12 months). The control group would receive TAU and be monitored using EMA.

Ethics and dissemination: This study has been approved by the Ethics Committee of the University Hospital Fundación Jiménez Díaz. It is expected that, in the near future, the mobile applications MEmind and eB2 can be implemented in routine clinical practice. Results will be disseminated through peer-reviewed journals and psychiatric congresses.

DETAILED DESCRIPTION:
Introduction: Over 800,000 die every year by suicide, while suicide attempts are estimated to be 20 times more frequent. Suicidal ideation (SI) is estimated to affect 2% of the population. Suicidal thoughts and behaviours (STB) increase the risk of death by suicide, impair people's quality of life and result in high healthcare costs.

New technologies can help us in the management and prevention of STB. Among other advantages, these devices open the possibility of implementing smartphone-based real-time monitoring. There are two main types of smartphone-based monitoring: active and passive. The active mode is also known as Ecological Momentary Assessment (EMA). EMA involves asking daily questions, resulting in real-time responses in the patient's usual environment. EMA provides a more accurate picture of the emotional and cognitive context in which SI appears, offering us the opportunity to identify its immediate predictors.

Passive monitoring -also called passive EMA- involves using the mobile phone's native sensors to collect information such as physical activity, mobility or sleep, which can be useful as proxy factors for mental state. The combination of active and passive monitoring produces valuable information to characterize people's behaviour, giving rise to what is known as an individual's digital phenotype (Barrigón et al., 2019). As it does not require patient effort, passive EMA can increase the acceptability of monitoring and counteract the so-called "EMA fatigue", which occurs when patients stop answering EMA questions.

A considerable number of studies have applied EMA technology to suicide research. In contrast, passive EMA has been used scarcely in suicidology.

A further step is to exploit EMA's potential to design digital therapeutic tools, providing continuous support in the patient's usual environment. This is known as Ecological Momentary Intervention (EMI). EMIs can be a useful add-on to traditional treatment, thanks to their 24-hour availability, low cost, and the possibility of continuing follow-up in a non-presential manner. Some studies have explored the effectiveness of EMI on suicidal behaviour, showing good acceptability and a reduction in SI after the intervention.

This is an up-and-coming area that may contribute to suicide prevention, which has not yet received sufficient attention in the scientific literature.

The SmartCrisis 2.0 randomized clinical trial aims to evaluate the effectiveness of an Ecological Momentary Intervention (EMI) combined with smartphone-based monitoring for the prevention of STB in patients at high risk of suicide.

Our hypotheses are as follows:

1. Before/after comparison: In the intervention group, there will be a significant reduction in STB and an improvement in functionality and quality of life after the follow-up period.
2. Comparison with control group: The intervention group will have a greater reduction in STB and a greater improvement in functioning and quality of life than the control group.
3. Feasibility and acceptability: The use of the eB2 and MEmind mobile applications will be feasible and well accepted by psychiatric patients.

Methods and analysis: Our sample will consist of patients with a history of recent STB treated at either one of these five locations: University Hospital Fundación Jiménez Díaz (Madrid, Spain), Rey Juan Carlos Hospital (Móstoles, Spain), and General Hospital of Villalba (Villalba, Spain), Centre hospitalier universitaire Montpellier (Montpellier, France) or Nîmes University Hospital (Nîmes, France).

Sample size calculation was performed using G*Power software, version 3.1. Based on previous clinical trials exploring the ability of crisis management interventions to reduce SI in the mid-term (Ducasse et al., 2018), the investigators estimated a target sample size enough to have 80% power to detect between-group differences of 6-7 points on the Columbia Suicide Severity Rating Scale (25% decrease in the intensity of SI in the intervention group). The alpha error was set at 5% and the power at 80%. A dropout rate of 20% and a randomization imbalance of 10% were assummed. With these settings, the investigators estimated that a total of 220 participants, 110 in each arm, were needed.

Before starting the clinical trial, a pilot will be conducted, in approximately 40 patients will be recruited. All of them will receive the SmartSafe EMI and be monitored using active and passive EMA. These patients will not be part of the final analysis. After three months of follow-up, when all participants have had time to try out the application, a focus group will be held between the research team, the attending clinicians and the patients in order to get their opinion on the intervention and to identify possible technical and human failures that could be improved before starting the clinical trial.

Once the clinical trial recruitment starts, attending psychiatrists will check their patients' eligibility during their regular appointment, explain the project in detail and invite them to participate. If patients agree to participate, they will be asked to sign the informed consent, after which they will be randomly assigned to the intervention group (EMI + EMA + TAU) or the control group (EMA + TAU).

At the baseline interview, a psychiatrist will assess the characteristics of the last suicidal event using the Brief Suicide Protocol, which has been previously published, and they will set up the SmartSafe intervention according to the patient's preferences. Next, a trained research assistant, blind to the patient's assigned arm, will administer the standardized questionnaires detailed below.

Patients will be followed for one year, with face-to-face visits at six months and one year. The attending psychiatrist will also check for STB using the Columbia Suicide Severity Rating Scale (CSSRS) at the 4th week, 11th week and 9th-month appointments. If participants cannot attend the follow-up visits, the assessments will be performed by phone. All questionnaires will be completed via the MEmind website.

The piloting is expected to take place between June and December 2021. Recruitment is expected to commence in January 2022 and to be completed by June 2023. Data collection will take place from 2022 to 2024. Data analysis will take place from 2022 to 2024. The investigators expect to publish partial results by the end of 2022 and final results by early 2025.

Digital monitoring will be performed using EMA. Two EMA modalities will be used: active using the MEmind app, and passive using the eB2 app.

The MEmind app asks short daily questions that appear on the mobile screen. Each day, 2-4 random questions will be asked at random times (respecting sleep hours) from the pool of 34 questions that make up the questionnaire based on the Salzburg Suicide Questionnaire.

The EMA questions belong to 6 categories:

* Suicidality (5 questions)
* Non-suicidal self injury (2 questions)
* Affect (9 questions)
* Interpersonal experiences (11 questions)
* Sleep (4 questions)
* Eating (3 questions) The eB2 app runs in the background and does not require user intervention. It collects real-time information from the patient's mobile phone (location, mobility, smartphone usage and sleep), stores it and downloads it to a server. All the information collected from the phone is transformed with a hash function. This hash function makes it impossible to know the original data but allows the analysis of behavioral patterns.

In addition to the smartphone-based monitoring, another digital assessment will be carried out: a neuropsychological assessment using a previously validated Virtual Reality environment, the "Spheres & Shield Maze Task". This tool recreates a maze with different tasks to assess decision-making, impulsivity, attention and cognitive inhibition.

Non-digital assessments will be carried out by attending psychiatrists and research assistants, all of them previously trained. All questionnaires will be completed on the MEmind website, which allows for easy completion and immediate uploading to databases.

Some of the main tools used will be the following:

* The Brief Suicide Questionnaire (BSQ) will be used to characterize the index event that motivated inclusion in the study (suicide attempt or emergency referral for SI). It includes questions on lethality, method and surrounding circumstances of the attempt, and lifetime history of suicidal behaviour.
* The CSSRS scale will be used to measure STB, both at baseline and follow-up visits.
* The investigators will verify suicide attempts and deaths by suicide through our organization's digital medical records, called the Casiopea software, which integrates information on ER visits, hospitalizations, and visits to specialist consultations. If a patient cannot be located, and there is no information in their record, the investigators will contact the patient's family telephone number. The investigators will also request access to the Spanish register of deaths and causes of death of the "Instituto Nacional de Estadística" [National Statistics Institute].

At the six-month follow-up visit, patients will complete a qualitative satisfaction survey with the following questions referring to each of the applications used (MEmind and eB2) and the face-to-face assessments.

Traditional statistical analyses will be performed using SPSS 24.0 statistical software. To compare SI at baseline with SI at the end of follow-up (CSSRS score), paired samples t-tests will be used. To compare the improvement in SI after follow-up between the intervention group and the control group, an independent samples t-test will be used.

Survival curves (time to a new suicidal event) will be calculated using the Kaplan-Meier test. The intervention group's survival curves and the control group will be compared using the log rank test. To assess the project's feasibility, participation rate, retention and percentage of EMA questions answered will be calculated.

Binary logistic regression will be used to explore the correlation between the study variables, obtaining crude and age- and sex-adjusted ORs. A multivariate regression model will also be built to assess the unique strength of the association of the variables. Cox regression analysis will be performed to explore variables associated with survival time (time until next event). All tests will be two-tailed, with a significance level of p<0.05 and 95% confidence intervals.

In addition to the traditional analyses, with the Signal Theory Department of the Carlos III University's support, unsupervised analyses will be carried out using machine learning techniques to create behavioral models and patient activity profiles.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a SA or an emergency referral for SI in the past month.
* Being able to understand and sign the informed consent form.
* Being fluent in Spanish
* Owning a smartphone with internet access and iOS or Android operating system.

Exclusion Criteria:

* Refusal to install the mobile application
* Inability to understand and sign the informed consent form for any reason.
* Institutionalized or incarcerated patients, without access to regular mobile phone use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of suicidal ideation | 6 months
  Our primary outcome will be reduction of suicidal ideation, measured at follow-up using the Columbia Suicide Severity Rating Scale
Reduction of suicidal ideation | 1 year
  Our primary outcome will be reduction of suicidal ideation, measured at follow-up using the Columbia Suicide Severity Rating Scale

SECONDARY OUTCOMES:
Acceptability of the mobile health applications | 6 months
  Acceptability of the mobile health applications measured by user satisfaction using satisfaction surveys
Acceptability of the mobile health applications | 1 year
  Acceptability of the mobile health applications measured by user satisfaction using satisfaction surveys
Feasibility of the project: Compliance | 6 months
  Feasibility measured by compliance with EMA questions (% of questions answered)
Feasibility of the project: Compliance | 1 year
  Feasibility measured by compliance with EMA questions (% of questions answered)
Feasibility of the project: Participation | 1 year
  Feasibility measured by participation rate (% of patients that accept to be enrolled in the project out of those invited to participate)
Feasibility of the project: Retention | 1 year
  Feasibility measured by retention rate (% of patients that remain in the study when the follow-up period is completed)
Reduction of suicide attempts | 6 months
  Reduction in the occurrence of suicide attempts registered as a clinical event (attended in the emergency room verified through the electronical clnical record)
Reduction of suicide attempts | 1 year
  Reduction in the occurrence of suicide attempts registered as a clinical event (attended in the emergency room verified through the electronical clnical record)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Barrigon, PhD, Principal Investigator — Instituto de Investigación Fundación Jiménez Díaz
Locations (1):
- Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrigon ML, Courtet P, Oquendo M, Baca-Garcia E. Precision Medicine and Suicide: an Opportunity for Digital Health. Curr Psychiatry Rep. 2019 Nov 28;21(12):131. doi: 10.1007/s11920-019-1119-8. PMID 31776806
- [Background] Berrouiguet S, Alavi Z, Vaiva G, Courtet P, Baca-Garcia E, Vidailhet P, Gravey M, Guillodo E, Brandt S, Walter M. SIAM (Suicide intervention assisted by messages): the development of a post-acute crisis text messaging outreach for suicide prevention. BMC Psychiatry. 2014 Nov 18;14:294. doi: 10.1186/s12888-014-0294-8. PMID 25404215
- [Background] Borges G, Nock MK, Haro Abad JM, Hwang I, Sampson NA, Alonso J, Andrade LH, Angermeyer MC, Beautrais A, Bromet E, Bruffaerts R, de Girolamo G, Florescu S, Gureje O, Hu C, Karam EG, Kovess-Masfety V, Lee S, Levinson D, Medina-Mora ME, Ormel J, Posada-Villa J, Sagar R, Tomov T, Uda H, Williams DR, Kessler RC. Twelve-month prevalence of and risk factors for suicide attempts in the World Health Organization World Mental Health Surveys. J Clin Psychiatry. 2010 Dec;71(12):1617-28. doi: 10.4088/JCP.08m04967blu. Epub 2010 Aug 24. PMID 20816034
- [Background] Bostwick JM, Pabbati C, Geske JR, McKean AJ. Suicide Attempt as a Risk Factor for Completed Suicide: Even More Lethal Than We Knew. Am J Psychiatry. 2016 Nov 1;173(11):1094-1100. doi: 10.1176/appi.ajp.2016.15070854. Epub 2016 Aug 13. PMID 27523496
- [Background] Czyz EK, Horwitz AG, Arango A, King CA. Short-term change and prediction of suicidal ideation among adolescents: a daily diary study following psychiatric hospitalization. J Child Psychol Psychiatry. 2019 Jul;60(7):732-741. doi: 10.1111/jcpp.12974. Epub 2018 Sep 24. PMID 30246870
- [Background] Davidson CL, Anestis MD, Gutierrez PM. Ecological Momentary Assessment is a Neglected Methodology in Suicidology. Arch Suicide Res. 2017 Jan 2;21(1):1-11. doi: 10.1080/13811118.2015.1004482. Epub 2016 Jan 29. PMID 26821811
- [Background] Ford-Gilboe M, Varcoe C, Scott-Storey K, Wuest J, Case J, Currie LM, Glass N, Hodgins M, MacMillan H, Perrin N, Wathen CN. A tailored online safety and health intervention for women experiencing intimate partner violence: the iCAN Plan 4 Safety randomized controlled trial protocol. BMC Public Health. 2017 Mar 21;17(1):273. doi: 10.1186/s12889-017-4143-9. PMID 28327116
- [Background] Franklin JC, Ribeiro JD, Fox KR, Bentley KH, Kleiman EM, Huang X, Musacchio KM, Jaroszewski AC, Chang BP, Nock MK. Risk factors for suicidal thoughts and behaviors: A meta-analysis of 50 years of research. Psychol Bull. 2017 Feb;143(2):187-232. doi: 10.1037/bul0000084. Epub 2016 Nov 14. PMID 27841450
- [Background] Ghanbari B, Malakouti SK, Nojomi M, Alavi K, Khaleghparast S. Suicide Prevention and Follow-Up Services: A Narrative Review. Glob J Health Sci. 2015 Sep 28;8(5):145-53. doi: 10.5539/gjhs.v8n5p145. PMID 26652085
- [Background] Hallensleben N, Glaesmer H, Forkmann T, Rath D, Strauss M, Kersting A, Spangenberg L. Predicting suicidal ideation by interpersonal variables, hopelessness and depression in real-time. An ecological momentary assessment study in psychiatric inpatients with depression. Eur Psychiatry. 2019 Feb;56:43-50. doi: 10.1016/j.eurpsy.2018.11.003. Epub 2018 Dec 5. PMID 30530103
- [Background] Kawohl W, Nordt C. COVID-19, unemployment, and suicide. Lancet Psychiatry. 2020 May;7(5):389-390. doi: 10.1016/S2215-0366(20)30141-3. No abstract available. PMID 32353269
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kleiman EM, Coppersmith DDL, Millner AJ, Franz PJ, Fox KR, Nock MK. Are suicidal thoughts reinforcing? A preliminary real-time monitoring study on the potential affect regulation function of suicidal thinking. J Affect Disord. 2018 May;232:122-126. doi: 10.1016/j.jad.2018.02.033. Epub 2018 Feb 17. PMID 29481996
- [Background] Kleiman EM, Turner BJ, Fedor S, Beale EE, Picard RW, Huffman JC, Nock MK. Digital phenotyping of suicidal thoughts. Depress Anxiety. 2018 Jul;35(7):601-608. doi: 10.1002/da.22730. Epub 2018 Apr 10. PMID 29637663
- [Background] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Background] Nordentoft M, Erlangsen A. Suicide-turning the tide. Science. 2019 Aug 23;365(6455):725. doi: 10.1126/science.aaz1568. No abstract available. PMID 31439766
- [Background] O'Connor RC, Portzky G. Looking to the Future: A Synthesis of New Developments and Challenges in Suicide Research and Prevention. Front Psychol. 2018 Nov 27;9:2139. doi: 10.3389/fpsyg.2018.02139. eCollection 2018. PMID 30538647
- [Background] Oquendo MA, Galfalvy HC, Choo TH, Kandlur R, Burke AK, Sublette ME, Miller JM, Mann JJ, Stanley BH. Highly variable suicidal ideation: a phenotypic marker for stress induced suicide risk. Mol Psychiatry. 2021 Sep;26(9):5079-5086. doi: 10.1038/s41380-020-0819-0. Epub 2020 Jun 23. PMID 32576966
- [Background] Porras-Segovia A, Molina-Madueno RM, Berrouiguet S, Lopez-Castroman J, Barrigon ML, Perez-Rodriguez MS, Marco JH, Diaz-Olivan I, de Leon S, Courtet P, Artes-Rodriguez A, Baca-Garcia E. Smartphone-based ecological momentary assessment (EMA) in psychiatric patients and student controls: A real-world feasibility study. J Affect Disord. 2020 Sep 1;274:733-741. doi: 10.1016/j.jad.2020.05.067. Epub 2020 May 26. PMID 32664009
- [Background] Reger MA, Stanley IH, Joiner TE. Suicide Mortality and Coronavirus Disease 2019-A Perfect Storm? JAMA Psychiatry. 2020 Nov 1;77(11):1093-1094. doi: 10.1001/jamapsychiatry.2020.1060. No abstract available. PMID 32275300
- [Background] Seppala J, De Vita I, Jamsa T, Miettunen J, Isohanni M, Rubinstein K, Feldman Y, Grasa E, Corripio I, Berdun J, D'Amico E; M-RESIST Group; Bulgheroni M. Mobile Phone and Wearable Sensor-Based mHealth Approaches for Psychiatric Disorders and Symptoms: Systematic Review. JMIR Ment Health. 2019 Feb 20;6(2):e9819. doi: 10.2196/mental.9819. PMID 30785404
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Smith KE, Juarascio A. From Ecological Momentary Assessment (EMA) to Ecological Momentary Intervention (EMI): Past and Future Directions for Ambulatory Assessment and Interventions in Eating Disorders. Curr Psychiatry Rep. 2019 Jun 4;21(7):53. doi: 10.1007/s11920-019-1046-8. PMID 31161276
- [Background] Spangenberg L, Glaesmer H, Hallensleben N, Rath D, Forkmann T. (In)stability of Capability for Suicide in Psychiatric Inpatients: Longitudinal Assessment Using Ecological Momentary Assessments. Suicide Life Threat Behav. 2019 Dec;49(6):1560-1572. doi: 10.1111/sltb.12547. Epub 2019 Mar 4. PMID 30834576
- [Background] Stanley B, Brown GK. Safety planning intervention: a brief intervention to mitigate suicide risk. Cogn Behav Pract. 2012;19(2):256-64.
- [Background] Yang B, Lester D. Recalculating the economic cost of suicide. Death Stud. 2007 Apr;31(4):351-61. doi: 10.1080/07481180601187209. PMID 17378112
- [Derived] Barrigon ML, Porras-Segovia A, Courtet P, Lopez-Castroman J, Berrouiguet S, Perez-Rodriguez MM, Artes A; MEmind Study Group; Baca-Garcia E. Smartphone-based Ecological Momentary Intervention for secondary prevention of suicidal thoughts and behaviour: protocol for the SmartCrisis V.2.0 randomised clinical trial. BMJ Open. 2022 Sep 20;12(9):e051807. doi: 10.1136/bmjopen-2021-051807. PMID 36127081